CLINICAL TRIAL: NCT06365918
Title: Phase I Study of VG2025 Delivered Intraperitoneally in Patients With Advanced Solid Tumors With Carcinomatosis
Brief Title: Study of VG2025 Delivered Intraperitoneally in Patients With Advanced Solid Tumors With Carcinomatosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0836; NCI-2024-03236 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor; Carcinomatosis
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intraperitoneal VG2025 (Experimental): Participants will receive VG2025 intraperitoneally over about 5 minutes on Days 1-3 of each 21-day cycle. Participants will be watched for side effects for about 2 hours after each dose.
  Up to 3 dose levels of VG2025 will be tested. At least 3 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of VG2025 given intraperitoneally is found.
  Interventions: Drug: VG2025

INTERVENTIONS:
Drug: VG2025 — Given by Intraperitoneal

SUMMARY:
To find the recommended dose of the investigational drug VG2025 that can be given intraperitoneally (given directly into the abdominal cavity) to participants with advanced solid tumors.

DETAILED DESCRIPTION:
Primary Objectives

1. To assess safety and tolerability of VG2025 following IP administration
2. To determine the Maximum Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D) of IP VG2025

Secondary Objectives

1. To estimate progression free survival
2. To characterize the biodistribution or shedding profile of detectable VG2025 DNA in tumor (biopsy samples), IP fluid, and blood
3. To evaluate IL-12, IL-15, and other cytokine levels in tumor (biopsy samples), IP fluid, and blood
4. To evaluate tumor CEA expression
5. To evaluate the objective response rate (ORR) and clinical benefit rate (CBR) of IP administration of VG2025 in the overall patient population and by dose level
6. To characterize changes in the IP and tumor immune microenvironment in response to treatment
7. To correlate circulating tumor DNA (ctDNA) with disease status

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
2. Pathology reviewed at MD Anderson Cancer Center.
3. Participants must have evidence of peritoneal carcinomatosis per imaging studies, as well as measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam.
4. Ability to understand and the willingness to sign a written informed consent document.
5. Age ≥ 18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
7. Had an interval of ≥ 4 weeks (28 days) since exposure to immunotherapy, an interval of ≥ 3 weeks (21 days) since exposure to systemic chemotherapy, an interval of ≥ 6 weeks (42 days) since exposure to nitrosourea, and an interval of ≥ 2 weeks (14 days) since exposure to radiotherapy, prior to dosing.
8. Participants must also:

   1. have either disease progression or intolerable toxicity after standard treatment.
   2. have received at least one prior line of systemic standard therapy.
   3. be fully recovered or at a grade 1 toxicity (based on CTCAE V5.0) due to prior chemotherapy, immunotherapy, or radiotherapy at Screening.
9. Participants must have adequate organ and marrow functions as defined below:

   1. Hemoglobin ≥ 80 grams (g)/liter (L).
   2. ANC ≥ 1.0 x 10^9/L.
   3. Lymphocyte count ≥ 0.75 x 109/L.
   4. Platelet count ≥ 100 x 109/L.
   5. Serum creatinine .1.5 x the upper limit of the reference range or Estimated Glomerular Filtration Rate (eGFR by Cockcroft-Gault formula) .45mL/min/1.73m2, for subjects with creatinine levels above institutional normal.
   6. Serum bilirubin ≤ 1.5 x the upper limit of the reference range.
   7. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x the upper limit of the reference range, or <5.0 x the upper limit of the reference range for participants with liver metastases.
   8. international normalization ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN, unless the participant is receiving anticoagulant therapy, in which case PT and partial thromboplastin time (PTT)/activated PTT (aPTT) must be within therapeutic range of intended use of anticoagulants.
   9. PTT or aPTT ≤ 1.5 x ULN unless the participant is receiving anticoagulant therapy as long as PT and PTT/aPTT is within therapeutic range of intended use of anticoagulants.
   10. pRBC transfusion is allowed as long as there is no active bleeding, but support for ANC and platelets are not allowed within 2 weeks of trial therapy initiation.
10. Participants whose baseline pulse oximetry is at least 90% on Room air.
11. The effects of VG2025 on the developing human fetus are unknown. For this reason and because Class II agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the participant presents with an applicable exclusionary factor which may be one of the following:

    * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
    * History of hysterectomy or bilateral salpingo-oophorectomy.
    * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
    * History of bilateral tubal ligation or another surgical sterilization procedure.

      * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Participant/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
      * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of VG2025 administration.
12. Females of childbearing potential must have a negative pregnancy test at Screening and on Day 1.
13. Willing to undergo intraperitoneal port placement and scheduled peritoneal fluid and peripheral blood draws, as well as pre- and on-treatment biopsies.
14. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
15. Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
16. Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
17. Participants with asymptomatic, new or progressive brain metastases (active brain metastases), except leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
18. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
19. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.

Exclusion Criteria:

1. Participants who are receiving any other investigational agents.

   • Participation in any previous trial when the last dose of the investigational agent was received within the last 4 weeks prior to dosing. If the half-life of the investigational drug was less than 5 days, participants may participate in the study sooner after 5 half-lives.
2. Participants with any primary CNS malignancy including glioma, or symptomatic and progressing CNS malignant lesions, including leptomeningeal disease are excluded. Participants with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging ([MRI or CT scan) during the screening period and off systemic steroids (for at least 2 weeks prior to first dose of VG2025).
3. Major surgery within 21 days prior to Screening commencement. Procedures such as Pleural drainage, tumor needle biopsy, feeding tube placement and central venous catheter are not considered major surgery.
4. Intercurrent serious infections within 28 days prior to Screening or treated systematically with intravenous antibiotics within 14 days prior to Screening.
5. Life-threatening illness unrelated to cancer.
6. Active Herpes infection.
7. Treatment with antiviral agents within 14 days prior to Screening commencement.
8. Known contraindications or hypersensitivity to the excipients of VG2025.
9. Participants with congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), unstable angina, serious uncontrolled cardiac arrhythmia, a myocardial infarction within 6 months prior to study entry or a history of myocarditis.
10. Known to test positive for human immunodeficiency virus (HIV), hepatitis B or C virus, or syphilis.

    For participants with positive test results of HIV that meet all the following eligibility criteria may be enrolled:
    * Have a T-cell (CD4+) count ≥ 350 cells/uL.
    * No History of opportunistic infections or other malignancies.
    * Have an HIV viral load less than 400 copies/mL prior to enrollment.
    * In the opinion of the investigator, their antiretroviral therapy (ART) or other HIV treatments will not interfere with the activity of the investigational product or cause any confusion with the assessment of the investigational drug toxicities.

    For participants with positive test results of HBV or HCV:

    -Participants with current active HBV or HCV infection or those with a history of HBV or HCV infection that are still on treatment are excluded. Participants with a past history of HBV and HCV infection are only allowed to participate, if they have a negative viral load test (HBV DNA Polymerase Chain Reaction (PCR) and HCV RNA PCR) within 30 days before screening.
11. Participants with a condition requiring systemic treatment with either corticosteroids (>10 milligrams (mg) daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to dosing. Inhaled or topical steroids, and adrenal replacement steroid doses, are permitted in the absence of active autoimmune disease.
12. Participants with active or documented history of autoimmune disease within 2 years prior to Screening commencement.

    Please note that subjects with vitiligo, resolved childhood asthma/atopy, autoimmune endocrinopathy on stable replacement therapy, or psoriasis not requiring systemic treatment within the past 2 years will be allowed.
13. Participants with history of primary immune deficiency.
14. Participants with history of organ transplant that requires use of immunosuppressive medications.
15. Use of any vaccines within 4 weeks prior to dosing.
16. Participants with any prior ≥ Grade 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE Grade >1 (as per NCI CTCAE Version 5.0).
17. Participants with any >Grade 1 toxicity (as per NCI CTCAE Version 5.0) related to prior anti-cancer therapy, except those that are deemed not clinically significant by the Investigator in discussion with the Clinical Trial Safety Manager.
18. Participants with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction, bleeding tendency), that would compromise the subject's ability to tolerate protocol therapy or would likely interfere with the study procedures or results.
19. Participants with history of prior HSV-1 encephalitis or encephalitis due to other etiology.
20. Participants with active infection causing fever (temperature > 38.1°C) or participants with unexplained fever (temperature > 38.1°C) within 7 days prior to the day of investigational product administration.
21. History of peritonitis, episode of inflammatory bowel disease, or diverticulitis within 6 months of enrollment.
22. Medical or surgical history that in the treating physician's opinion would make the subject not a suitable candidate for IP therapy. Examples would include surgically documented extensive intraperitoneal adhesions or large volume ascites that requires therapeutic paracentesis within the last 2 weeks.
23. Any other illnesses/conditions that in the investigator's opinion would adversely affect the safety of oncolytic virus therapy.
24. Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
25. Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
26. History of allergic reactions attributed to compounds of similar chemical or biologic composition to VG2025, or other agents used in study.
27. Concomitant medications or substances that have the potential to affect the activity or pharmacokinetics of the study agent(s): anti-viral agents, and immunosuppressive agents.
28. Participants with psychiatric illness/social situations that would limit compliance with study requirements.
29. Pregnant women are excluded from this study because VG2025 is Class II agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with VG2025, breastfeeding should be discontinued if the mother is treated with VG2025. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org